CLINICAL TRIAL: NCT02241369
Title: A Study of HPV Specific Immunotherapy in Subjects With HPV6 Associated Aerodigestive Precancerous Lesions and Malignancies
Brief Title: Immunotherapy in Subjects With HPV-6 Associated Aerodigestive Precancerous Lesions and Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPV-006
Record Dates: First submitted 2014-09-11; First posted 2014-09-16 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Aerodigestive Precancerous Lesions and Malignancies
Keywords: Aerodigestive Lesions and Malignancies; Human Papillomavirus; Squamous Cell Carcinoma
MeSH Terms: conditions — Neoplasms; Carcinoma, Squamous Cell | interventions — rocakinogene sifuplasmid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort I (Experimental): 3 mg of INO-3106 (D0); 6 mg of INO-3106 (Wk3); 6 mg of INO-3106 + 1 mg of INO-9012 (Wk6); 6 mg of INO-3106 + 1 mg of INO-9012 (Wk9);
  Interventions: Biological: INO-3106, INO-9012
- Cohort II (Experimental): 6 mg of INO-3106 in combination with 1 mg of INO-9012, or at the MTD determined above at D0, Wk3, Wk6, Wk9
  Interventions: Biological: INO-3106, INO-9012

INTERVENTIONS:
Biological: INO-3106, INO-9012

SUMMARY:
This is a Phase I, open-label study to evaluate the safety, tolerability, and immunogenicity of INO-3106 alone or in combination with INO-9012 DNA vaccines delivered by Electroporation to subjects with HPV6 associated aerodigestive precancerous lesions and malignancies.

DETAILED DESCRIPTION:
This is a Phase I, open-label, study to evaluate the safety, tolerability, and immunogenicity of 3 mg or 6 mg INO-3106 alone or in combination with 1 mg of INO-9012 (DNA plasmid encoding human interleukin 12) delivered by electroporation (EP) in subjects with HPV6 associated aerodigestive precancerous lesions and malignancies. Subjects will be enrolled in 2 cohorts (3 subjects in each cohort):

Cohort I: First 3 subjects will be enrolled sequentially and will receive INO-3106 alone or in combination with INO-9012.

Cohort II: The next 3 subjects will be treated with 6 mg of INO-3106 and 1 mg of INO-9012, or at the MTD (Maximum Tolerated Dose) determined in Cohort I.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written Ethics Committee approved informed consent
* Age ≥18 years
* Histologically documented HPV-6 positive aerodigestive invasive malignancy (mucosal squamous cell head and neck cancer or lung cancer) who have completed therapies such as radiation/chemoradiation/chemotherapy; or
* Histologically documented HPV-6 positive papilloma or HPV-6 related premalignant lesion (i.e., carcinoma in situ) in aerodigestive or head and neck regions.
* Prior to study entry, subjects will have exhausted all treatments that are/have been used in these indications which may include any combination of surgery, anti-viral therapy, chemotherapy and/or radiation therapy.
* Core biopsy must be obtained prior to enrollment to confirm invasive cancer. Archival material is allowed.
* Adequate bone marrow, hepatic, and renal function. ANC (Absolute Neutrophil Count) ≥ 1.5x109 cell/ml, platelets ≥75,000 cells/mm3, hemoglobin ≥ 9.0 g/dL, concentrations of total serum bilirubin within 1.5 x upper limit of normal (ULN), AST, ALT within 2.5x ULN, CPK within 2.5 x ULN, serum creatinine ≤ 1.5x ULN
* ECOG (Eastern Cooperative Oncology Group) performance status of 0-2

Exclusion Criteria:

* Participation in a clinical trial within 30 days before entry
* Any cardiac pre-excitation syndromes, e.g. Wolff-Parkinson-White syndrome
* Presence of metal implants within 5 cm of the planned site(s) of injection
* Anticipated concomitant immunosuppressive therapy (excluding non-systemic inhaled, topical skin and/or eye drop-containing corticosteroids)
* Administration of any vaccine within 6 weeks of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-05; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Adverse events measured and graded in accordance with "Common Terminology Criteria for Adverse Events (CTCAE)", NCI version 4.03 | Up to 6 months
Injection site reactions including skin erythema, induration pain and tenderness at administration site | Up to 15 weeks

SECONDARY OUTCOMES:
HPV6 specific Ig levels | Up to 6 months
Number of antigen-specific IFN-γ-secreting cells in response to stimulation with HPV6 by antigen-specific IFN-γ ELISpot assays | Up to 6 months
Cytotoxic T cells in response to HPV6 specific immunotherapy by flow cytometry | Up to 6 months

OTHER OUTCOMES:
Time to new anti-cancer therapy | First dose to Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Skolnik, MD, Study Director — Inovio Pharmaceuticals
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor's Website — http://www.inovio.com